CLINICAL TRIAL: NCT07138807
Title: Comparative Effectiveness of Muscle Energy Technique and Neck Calliet Exercises on Mechanical Neck Pain and Disability Due to Trapezius Trigger Point Among Nurses
Brief Title: Effect of MET vs Neck Calliet Exercises on Neck Pain and Disability in Nurses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Fiza Tariq, Clinical Research Investigator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MET_Calliet_NeckPain_Nurses
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: MET, Neck Calliet Exercise, Cervical ROM, VAS, NDI
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MET Group (Experimental): Participants received Muscle Energy Techniques (MET) for 4 weeks, 3 sessions per week, in addition to TENS
  Interventions: Behavioral: Muscle Energy Technique
- Calliet Exercise Group (Experimental): Participants performed Neck Calliet Exercises for 4 weeks, 3 sessions per week, in addition to TENS.
  Interventions: Other: Neck Calliet exercise

INTERVENTIONS:
Behavioral: Muscle Energy Technique — Participants in this group received Muscle Energy Techniques targeting the upper trapezius trigger points. Treatment was provided 3 sessions per week for 4 weeks. Each session included post-isometric relaxation techniques with stretching, along with baseline TENS therapy.Participants performed Neck Calliet Exercises focusing on cervical flexion, extension, rotation, and lateral flexion. Exercises were done under supervision, 3 times per week for 4 weeks. All participants also received baseline TENS therapy.
  Arms: MET Group
Other: Neck Calliet exercise — Neck Calliet exercise
  Arms: Calliet Exercise Group

SUMMARY:
This study compares the effectiveness of Muscle Energy Techniques (MET) and Neck Calliet Exercises in managing mechanical neck pain and associated disability due to trapezius trigger points among nurses. A total of 38 female nurses were randomly assigned to two intervention groups, each receiving therapy for four weeks. Pain, cervical range of motion, and disability outcomes were assessed.

DETAILED DESCRIPTION:
Musculoskeletal disorders, particularly neck pain, are highly prevalent among nurses due to repetitive strain, prolonged standing, and non-ergonomic work postures. One of the major contributors to mechanical neck pain is the presence of active myofascial trigger points in the trapezius muscle, which limit cervical range of motion (CROM) and increase disability.This single-blinded, randomized clinical trial aimed to compare the effectiveness of Muscle Energy Techniques (MET) and Neck Calliet Exercises in reducing mechanical neck pain and disability among nurses with trapezius trigger points. Thirty-eight participants were randomly divided into two groups: Group A received MET, and Group B performed Neck Calliet Exercises. Both groups also received TENS (Transcutaneous Electrical Nerve Stimulation) therapy as a baseline treatment. Each participant received treatment three times per week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female nurses
* Between 18 and 30 years of age
* Having mechanical neck discomfort that is confined to the cervical or bilateral scapular regions (pain level must be 3-5 VAS)
* There must be at least one trigger point in trapezius muscle
* The participant must be ready to participate No clinical therapy for neck pain must have been performed in the preceding month

Exclusion Criteria:

* A recent medical history including surgery on the shoulder or neck
* Signs of myelopathy in the clinic or radiculopathy
* Diagnosed Fibromyalgia syndrome, psychiatric problems
* Pregnancy
* Cervical stenosis, malignancy (cervical, breast cancer)
* Thoracic outlet syndrome
* Vestibulobasilar artery syndrome
* Whiplash injury
* Diagnosis of migraine
* Diabetes type I, systematic illness of cardio-respiratory system
* Congenital deformities affecting the spine, shoulders, and limbs
* Osteoporosis of cervical spine or cervical myeloma

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female nurses aged 25 to 45 years with mechanical neck pain and active trapezius trigger points were included in the study. The gender restriction was applied to ensure sample homogeneity and to control for occupational and physiological factors that may influence the outcomes.
Enrollment: 38 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Pain Intensity Pain intensity | Baseline and 4 weeks
  Change in neck pain intensity was assessed using the Visual Analogue Scale (VAS), measured before and after 4 weeks of intervention.
Functional Disability | Baseline and 4 weeks
  Functional disability was evaluated using the Neck Disability Index (NDI) at baseline and after 4 weeks of treatment.

SECONDARY OUTCOMES:
Cervical Range of Motion | Baseline and 4 weeks
  Cervical range of motion (flexion, extension, rotation, lateral flexion) was measured using a universal goniometer pre- and post-intervention to assess changes in mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tanveer Ahmad, HOD Surgery, Principal Investigator — The University of Faisalabad
Locations (1):
- The University of Faisalabad, Faisalabad, Punjab Province, Pakistan